CLINICAL TRIAL: NCT02115802
Title: Local Field Potential Correlates of Motor Behavior and Pathological Signs in Movement Disorders for Development of Closed Loop Stimulation Systems
Brief Title: LFP Correlates of Movement Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colorado Neurological Institute (Other)
Collaborators: Swedish Medical Center (Other); Medtronic (Industry)
Responsible Party: Principal Investigator, Adam O Hebb, Principal Investigator, Colorado Neurological Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Activa PC+S
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Activa PC+S (Experimental): Specific features of LFP recorded from the deep brain nuclei will be examined for possible correlation with different natural behaviors, such as movement, walking, or speech.
  Interventions: Device: Activa PC+S

INTERVENTIONS:
Device: Activa PC+S — Subjects will undergo placement of bilateral standard Deep Brain Stimulation (DBS) electrodes (Medtronic model 3387/3389) and implantation of the Activa PC+S, a modified impulse generator (IPG) for DBS with the added technology of neural signal recording.

SUMMARY:
The purpose of this study is to record electrical brain activity during DBS surgery and after DBS surgery using the Medtronic Activa PC+S deep brain stimulation (DBS) system, a modified DBS pulse generator. The goal of the study is to investigate if the electrical brain activity can help customize DBS therapy.

DETAILED DESCRIPTION:
The Activa PC+S system will be implanted and programmed under the same clinical procedures and standard of care as the Activa PC system. After implantation and standard clinical programming, participants in our research study will be asked to return for additional research visits where the recording sub-circuit of the device will be activated and local field potentials (LFP) will be recorded in the device and transmitted through telemetry to a base station for storage and future analysis. The sensing, or recording, sub-circuit will be disabled, non-invasively, at the end of each research visit to minimize impact to battery life of the device.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants must be undergoing DBS lead placement for Parkinson's Disease that requires them to be awake during microelectrode recording.
* Potential participants have been treated with levodopa/carbidopa, and with a dopamine agonist, at the maximal tolerated doses as determined by a movement disorders neurologist.
* Potential participants must have a Hoehn and Yahr stage >= 2 in the medications OFF state.
* Potential participants must have documented improvement in motor signs on versus off dopaminergic medication, with a change in the Unified Parkinson's Disease Rating Scale motor (UPDRS III) score of >= 30% off to on medication. Patients with tremor predominant form of PD, quantified as a UPDRS tremor score in any one limb greater than or equal to 3 and UPDRS sum of axial score (speech, posture, gait, balance) less than or equal to 5, who do not reach the 30% threshold, may be included.
* Potential participants must have evidence of complications of medication, e.g., wearing off signs, fluctuating responses and/or dyskinesias, and/or medication refractory tremor, and/or impairment in the quality of life on or off medication.
* Potential participants must have the ability to understand instructions in English.
* Potential participants are males or females between the ages of 21 and 75.

Exclusion Criteria:

* Individuals who are pregnant, breastfeeding, or are capable of becoming pregnant and not using an acceptable method of birth control. Acceptable methods of birth control include hormonal contraceptives, intrauterine device, abstinence or spermicide and barrier.
* Individuals who have magnetic resonance imaging (MRI) scans demonstrating cortical atrophy out of proportion to age.
* Individuals who have MRI scans showing focal brain lesions that could indicate a nonidiopathic movement disorder.
* Individuals who have major comorbidity increasing the risk of surgery such as prior stroke, severe hypertension, severe diabetes, or need for chronic anticoagulation other than aspirin.
* Individuals who have had any prior intracranial surgery.
* Individuals who have clinically active depression defined according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria and scored on a validated depression assessment scale.
* Individuals who have significant cognitive impairment and/or dementia as determined by a standardized neuropsychological battery.
* Individuals who have a history of seizures.
* Individuals who are immunocompromised.
* Individuals who have an active infection.
* Individuals who require diathermy, electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS) to treat a chronic condition.
* Individuals who have an implanted electronic device such as a neurostimulator, cardiac pacemaker or medication pump.
* Individuals who, at the discretion of the research team member, lack the cognitive ability to understand the instructions and fully participate in research tasks.
* Unable to understand written and spoken instructions in English. Individuals who carry a concomitant diagnosis that would preclude them from fully participating in the research tasks due to difficulties associated with comprehending instructions, cooperating with research tasks, or otherwise rendering the individuals incapable of participating in the research tasks. Examples could include a visual or hearing impairment preventing the individual from viewing a computer screen or hearing instructions.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Specific features of local field potentials recorded from the deep brain nuclei during different natural behaviors, such as movement, walking, or speech. | 3 years
  The broadband time domain neural signal across all bipolar pairs will be recorded in series while subjects perform structured behavioral tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Adam O Hebb, MD, Principal Investigator — Colorado Neurological Institute
Locations (1):
- Colorado Neurological Institute, Englewood, Colorado, United States